CLINICAL TRIAL: NCT05035121
Title: Effects of Milk or Soy Milk Combined With Mild Resistance Exercise on the Muscle Mass and Muscle Strength in Very Old Nursing Home Residents With Sarcopenia
Brief Title: Effect of Nutrition Supplementation Combined With Resistance Exercise in Elderly With Sarcopenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Jiun-Rong Chen, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201702034
Record Dates: First submitted 2021-05-24; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Sarcopenia
Keywords: sarcopenia; milk; soy milk; resistance exercise
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The participants were divided into three groups, such as control, milk supplement and soy milk supplement. The milk and soy milk groups provided 200 mL milk or soy milk two times per day. Moreover, all participants joined the resistance exercise training program, three times per week (30min/time).
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- milk supplement (Experimental): The milk group provided 200 mL milk two times per day. The participants joined the resistance exercise training program, three times per week (30 min/time) during 12 weeks.
  Interventions: Dietary Supplement: milk supplement; Behavioral: resistance exercise
- soy milk supplement (Experimental): The soy milk group provided 200 mL soy milk two times per day. The participants joined the resistance exercise training program, three times per week (30 min/time) during 12 weeks.
  Interventions: Dietary Supplement: soy milk supplement; Behavioral: resistance exercise
- control (Placebo Comparator): The participants joined the resistance exercise training program, three times per week (30 min/time) during 12 weeks.
  Interventions: Behavioral: resistance exercise

INTERVENTIONS:
Dietary Supplement: milk supplement — Intervention groups provided 200 mL long life milk two times per day at morning and afternoon. The participants joined the resistance exercise training program, three times per week (30 min/time)
  Arms: milk supplement
Dietary Supplement: soy milk supplement — Intervention groups provided 200 mL long life soy milk two times per day at morning and afternoon. The participants joined the resistance exercise training program, three times per week (30 min/time)
  Arms: soy milk supplement
Behavioral: resistance exercise — The participants joined the resistance exercise training program, three times per week (30 min/time)

SUMMARY:
The purpose of this study was determine whether milk or soy milk supplements combined with resistance exercise improved sarcopenia in the elderly. This study was randomized controlled trail that recruited elderly people ≧65 years old with sarcopenia in the nursing home of Taipei Veterans General Hospital Su-Ao and Yuanshan Branch from June 2017 to December, 2017. The participants were divided into three groups, such as control, milk supplement and soy milk supplement. The milk and soy milk groups provided 200 mL milk or soy milk two times per day. Moreover, all participants joined the resistance exercise training program, three times per week (30 min/time). After 12 weeks, the anthropometry, sarcopenia index, blood biochemical index, nutrition status index, inflammation index, insulin resistance index, and dietary intake were measured.

DETAILED DESCRIPTION:
The anthropometry data included body weight and body fat. The sarcopenia index included appendicular skeletal muscle mass index, calf circumferences, hand grip and gait speed. Moreover, blood biochemical index (liver function as ALT, kidney function as creatinine), nutrition status index (prealbumin, 25-hydroxyvitamin D) were also analyzed. The blood hsCRP level was as inflammation index and insulin resistance index included fasting blood sugar, insulin, HbA1c and HOMA-IR. The daily dietary intake were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 65 years old
* No allergies to milk and soy milk
* Sarcopenia cases (AWGS)
* Active ability

Exclusion Criteria:

* End-of-life patient or estimated death within six months
* Last stage of cancer
* Chronic kidney disease stage 4

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
appendicular skeletal muscle mass in kilograms | baseline
  The appendicular skeletal muscle mass was evaluated by bioelectrical impedance (BIA) analysis (Inbody S10, Inbody Inc., Seoul, South Korea)
Change from baseline appendicular skeletal muscle mass at 6 weeks | 6 weeks
  The appendicular skeletal muscle mass was evaluated by bioelectrical impedance (BIA) analysis (Inbody S10, Inbody Inc., Seoul, South Korea)
Change from baseline appendicular skeletal muscle mass at 12 weeks | 12 weeks
  The appendicular skeletal muscle mass was evaluated by bioelectrical impedance (BIA) analysis (Inbody S10, Inbody Inc., Seoul, South Korea)
height in meters | baseline
  Height was measured by height meter
Change baseline weeks height at 6 weeks | 6 weeks
  Height was measured by height meter
Change from baseline height at 12 weeks | 12 weeks
  Height was measured by height meter
appendicular skeletal muscle mass index in kg/m^2 | baseline
  The appendicular skeletal muscle mass muscle mass and height was combined to report appendicular skeletal muscle mass index in kg/m^2.
Change from baseline appendicular skeletal muscle mass index at 6 weeks | 6 weeks
  The appendicular skeletal muscle mass muscle mass and height was combined to report appendicular skeletal muscle mass index in kg/m^2.
Change from baseline appendicular skeletal muscle mass index at 12 weeks | 12 weeks
  The appendicular skeletal muscle mass muscle mass and height was combined to report appendicular skeletal muscle mass index in kg/m^2.
calf circumferences in centimeter | baseline
  calf circumferences (cm) was measured by using a measuring tape to go around the thickest point of the calf and stick tightly without squeezing the skin.
Change from baseline calf circumferences at 6 weeks | 6 weeks
  calf circumferences (cm) was measured by using a measuring tape to go around the thickest point of the calf and stick tightly without squeezing the skin.
Change from baseline calf circumferences at 12 weeks | 12 weeks
  calf circumferences (cm) was measured by using a measuring tape to go around the thickest point of the calf and stick tightly without squeezing the skin.
hand grip in kilograms | baseline
  The muscle strength was evaluated with the hand-grip strength (kg) using a Smedley dynamometer (TTM-YD, Tsutsumi Industries, Tokyo, Japan)
Change from baseline hand grip at 6 weeks | 6 weeks
  The muscle strength was evaluated with the hand-grip strength (kg) using a Smedley dynamometer (TTM-YD, Tsutsumi Industries, Tokyo, Japan)
Change from baseline hand grip at 12 weeks | 12 weeks
  The muscle strength was evaluated with the hand-grip strength (kg) using a Smedley dynamometer (TTM-YD, Tsutsumi Industries, Tokyo, Japan)
gait speed in meter per second | baseline
  The gait speed test was performed by recording the average time of walking 6 meters and representing with the distance (m) per second.
Change from baseline gait speed at 6 weeks | 6 weeks
  The gait speed test was performed by recording the average time of walking 6 meters and representing with the distance (m) per second.
Change from baseline gait speed at 12 weeks | 12 weeks
  The gait speed test was performed by recording the average time of walking 6 meters and representing with the distance (m) per second.

SECONDARY OUTCOMES:
blood alanine transaminase activity in U/L | baseline
  The blood alanine transaminase (ALT) activity in U/L was measured as liver function index by automated clinical chemistry analyzer.
Change from baseline blood alanine transaminase activity at 12 weeks | 12 weeks
  The blood alanine transaminase (ALT) activity in U/L was measured as liver function index by automated clinical chemistry analyzer.
blood creatinine level in mg/dL | baseline
  The blood creatinine level was measured as kidney function by automated clinical chemistry analyzer.
Change from baseline blood creatinine level at 12 weeks | 12 weeks
  The blood creatinine level was measured as kidney function by automated clinical chemistry analyzer.
blood prealbumin level in mg/dL | baseline
  The blood prealbumin level in mg/dL as the index of nutritional status were measured by automated clinical chemistry analyzer.
Change from baseline blood prealbumin level at 12 weeks | 12 weeks
  The blood prealbumin level in mg/dL as the index of nutritional status were measured by automated clinical chemistry analyzer.
blood 25-hydroxyvitamin D level in ng/mL | baseline
  The blood 25-hydroxyvitamin D level in ng/mL as the index of nutritional status were measured by automated clinical chemistry analyzer.
Change from baseline blood 25-hydroxyvitamin D level at 12 weeks | 12 weeks
  The blood 25-hydroxyvitamin D level in ng/mL as the index of nutritional status were measured by automated clinical chemistry analyzer.
High sensitive C-reactive protein in mg/dL | baseline
  High sensitive C-reactive protein (hsCRP) as the inflammatory indicator were measured by automated clinical chemistry analyzer.
Change from baseline High sensitive C-reactive protein at 12 weeks | 12 weeks
  High sensitive C-reactive protein (hsCRP) as the inflammatory indicator were measured by automated clinical chemistry analyzer.
blood fasting blood sugar in mg/dL | baseline
  The blood fasting blood sugar level in mg/dL as the insulin resistance index was measured by automated clinical chemistry analyzer.
Change from baseline blood fasting blood sugar at 12 weeks | 12 weeks
  The blood fasting blood sugar level in mg/dL as the insulin resistance index was measured by automated clinical chemistry analyzer.
blood insulin level in milli-international unit/L | baseline
  The blood insulin level in milli-international unit/L as the insulin resistance index was measured by commercial kits.
Change from baseline blood insulin level at 12 weeks | 12 weeks
  The blood insulin level in milli-international unit/L as the insulin resistance index was measured by commercial kits.
blood HbA1c in percentage | baseline
  The blood HbA1c in percentage as the insulin resistance index was measured by automated clinical chemistry analyzer.
Change from baseline blood HbA1c at 12 weeks | 12 weeks
  The blood HbA1c in percentage as the insulin resistance index was measured by automated clinical chemistry analyzer.
Homeostasis model assessment-insulin resistance index (HOMA-IR) | baseline
  HOMA-IR was calculated according to the formula: fasting insulin (μU/mL) x fasting glucose (mmol/L)/22.5
Change from baseline homeostasis model assessment-insulin resistance index (HOMA-IR) at 12 weeks | 12 weeks
  HOMA-IR was calculated according to the formula: fasting insulin (μU/mL) x fasting glucose (mmol/L)/22.5
blood insulin-like growth factor 1 in mg/dL | baseline
  The blood insulin-like growth factor 1 (IGF-1) level considered to be related with the protein synthesis in muscle was measured by chemiluminescence immunoassay.
Change from baseline blood insulin-like growth factor 1 at 12 weeks | 12 weeks
  The blood insulin-like growth factor 1 (IGF-1) level considered to be related with the protein synthesis in muscle was measured by chemiluminescence immunoassay.

OTHER OUTCOMES:
diet assessment | baseline
  Dietary data were collected based on the meal menu of the nursing home including one weekday and two weekends at the beginning and the end of the experiment. Caregivers recorded the actual food intake by participants. The intake of total energy, carbohydrate, protein and fat was analyzed with E Kitchen Nutrients Analysis Software (E Kitchen Business, Taichung, Taiwan) based on the food and nutrient database created by the Organization Act of the Food and Drug Administration, Ministry of Health and Welfare, Taiwan.
Change from baseline diet assessment at 12 weeks | 12 weeks
  Dietary data were collected based on the meal menu of the nursing home including one weekday and two weekends at the beginning and the end of the experiment. Caregivers recorded the actual food intake by participants. The intake of total energy, carbohydrate, protein and fat was analyzed with E Kitchen Nutrients Analysis Software (E Kitchen Business, Taichung, Taiwan) based on the food and nutrient database created by the Organization Act of the Food and Drug Administration, Ministry of Health and Welfare, Taiwan.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, New Taipei City, Taiwan